CLINICAL TRIAL: NCT04250584
Title: Investigation of the Substantial Equivalence of a Novel Mandibular Advancement Device, iSlpr™, With SomnoDent® Classic, in a Non-inferiority Study, in the Treatment of Snoring and Mild to Moderate Obstructive Sleep Apnoea.
Brief Title: Substantial Equivalence of iSlpr™ and SomnoDent® Classic in the Treatment of Snoring and Mild to Moderate Sleep Apnoea.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BioAnalytics Holdings Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAH001
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Sleep Apnea; Snoring
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Device (Experimental): Novel Mandibular Advancement Device
  Interventions: Device: iSlpr™
- Predicate Device (Active Comparator): Predicate Mandibular Advancement Device
  Interventions: Device: SomnoDent® Classic

INTERVENTIONS:
Device: iSlpr™ — mandibular advancement device
  Arms: Test Device
Device: SomnoDent® Classic — mandibular advancement device
  Arms: Predicate Device

SUMMARY:
The study is a thirty three week, prospective, open-label, randomized, parallel-group non-inferiority study.

The study aims to investigate the Substantial Equivalence of a novel mandibular device called iSlpr™, produced by BioAnalytics, to a currently approved device, SomnoDent® Classic, in the treatment of mild to moderate Obstructive Sleep Apnoea (OSA) and snoring.

DETAILED DESCRIPTION:
The objective of this study is to determine if the BioAnalytics device, iSlpr™, has a similar safety and efficacy profile to a commonly used device, SomnoDent® Classic, in the treatment of snoring and mild to moderate Obstructive Sleep Apnoea.

The target population will be males and females aged from 18 years to less than 75 years, who have been diagnosed with snoring and mild to moderate sleep apnoea.

Participants will remain on study from screening visit to end of study visit; a total of approximately 33 weeks.

This study includes -

* a screening period of up to 28 days
* a 2 week device initiation period
* a 24 week treatment period

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and younger than 75 years at time of screening
* Snoring and mild to moderate sleep apnoea ( AHI > 5 and < 30 per hr)
* Written informed consent
* Able to complete the study procedures within the study timeline.

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Central sleep apnoea
* Severe respiratory disorders
* Loose teeth or advanced periodontal disease
* Lateral bruxers
* Full or partial dentures
* Temporomandibular Joint (TMJ) abnormalities, pain or dysfunction
* Other teeth, jaw or gum disorders would preclude use of the device
* Cardiovascular comorbidities or stroke/heart attack in past 12 months
* Drug-addiction
* Major Depressive Disorder or psychosis
* Undergoing concomitant therapy for OSA/Snoring
* current or previous therapy with SomnoDent Classic
* Professional drivers or machine operators required to be undertaking CPAP

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
AHI | 24 weeks
  Apnea Hypopnea Index
ODI | 24 weeks
  Oxygen Desaturation Index

IPD SHARING:
Plan to Share IPD: No